CLINICAL TRIAL: NCT06683625
Title: Effects of Intense Physical Exertion on Neurotransmitter Levels, Stress, and Recovery in Relation to Energy Availability in Athletes
Brief Title: Neurotransmitter Analysis, Stress, and Energy Availability in Athletes
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Joanna Ostapiuk-Karolczuk, PhD, Poznan University of Physical Education
Other Study IDs: RowersMF2024
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: neurotransmitters; low energy availability; athletes; fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Eight female athletes
  Interventions: Diagnostic Test: 6K Max Effort Erg Test
- Group 2: 19 male athletes
  Interventions: Diagnostic Test: 6K Max Effort Erg Test

INTERVENTIONS:
Diagnostic Test: 6K Max Effort Erg Test — "6K Max Effort Erg Test", involves participants completing a 6000-meter rowing distance on an ergometer as quickly as possible. This test is designed to measure peak endurance and performance under controlled conditions and will serve as a primary assessment of each athlete's physical output and adaptive capacity.

SUMMARY:
The goal of this observational study is to examine if there is a correlation between energy deficiency, neurotransmitter levels, and exercise test performance among athletes in the Polish national rowing team. The main questions it aims to answer are:

Does relative energy deficiency (RED) impact neurotransmitter levels and, consequently, athletic performance? Can monitoring energy availability, neurotransmitter levels, and psychological factors provide insights into physiological and psychological adaptations to intense training? Researchers will compare results obtained before the exercise test with those taken immediately after and following a 1-hour recovery period to assess changes in performance, biochemical markers, and psychological responses.

Participants will:

* Engage in a standardized exercise test.
* Undergo assessments of energy availability, neurotransmitter levels, and performance at multiple time points (pre-exercise, immediately post-exercise, and post-1-hour recovery).
* Complete psychological questionnaires assessing stress levels, recovery, and energy availability.

This study aims to identify potential links between energy status, biochemical responses, psychological well-being, and athletic performance, allowing for targeted interventions to optimize training outcomes.

DETAILED DESCRIPTION:
The primary goal of this project is to optimize athletic training for the national rowing team through comprehensive multi-dimensional monitoring. This approach aims to enhance athletes' performance capabilities and readiness for high-level competition. The Polish national rowing team consistently wins medals at international events, with the Olympic medal being the ultimate achievement for these athletes. Given this high standard, special attention is placed on preparing the athletes, not only in terms of physical readiness but also through continuous monitoring of adaptive processes. This proactive approach enables early detection of adverse changes, allowing for rapid adjustments to the training process to prevent fatigue and overtraining.

Building on the previous year's findings, this project focuses on the effects of relative energy deficiency (RED) in sports. Introduced by the International Olympic Committee in 2014, RED refers to a syndrome of impairments that arise from low energy availability (EA) due to an imbalance between energy intake and expenditure relative to lean body mass. In high-performance sports like rowing, athletes experience internal and external pressures to maintain peak performance, which often impacts energy intake and expenditure. Low energy availability (LEA) initially leads to negative energy balance and weight loss, as the body's energy reserves are used to meet demand. Over time, chronic LEA results in metabolic and physiological adaptations, reducing total energy expenditure to prevent further weight loss. While body weight and fat mass may stabilize, athletes can experience compromised physiological functions due to LEA.

LEA impacts recovery, muscle mass, neuromuscular function, and increases injury risk, all of which can detrimentally affect performance. Sustained LEA aimed at reducing body mass or fat levels can lead to health and performance declines, a pattern seen in both male and female athletes. Recent awareness highlights that male rowers, previously assumed to be protected due to their higher lean mass and body size, may also experience RED-S. The demands of high-level rowing, often involving six hours of intense daily training with long endurance sessions and strength workouts, create challenges in meeting energy requirements.

This project involves biochemical assessments alongside psychological questionnaires to monitor athletes' stress, recovery, and energy availability. Such comprehensive monitoring provides insights into both the physical and mental responses to training stressors, supporting the development of tailored interventions for optimal performance and health in elite rowers.

ELIGIBILITY:
Inclusion Criteria:

* Gender and Biological Sex Alignment: Participants' self-identified gender must align with their biological sex due to the effects of sexual dimorphism on athletic performance.

Sex: Both male and female athletes are eligible to participate. Training Level: Participants must be highly trained, with a minimum of 5 years of consistent, high-level athletic training experience.

Experience: Participants should have competitive experience at a regional, national, or international level.

Health Status: Participants must be healthy, with no current or chronic medical conditions, injuries, or diseases that could affect study outcomes.

Exclusion Criteria:

* Gender-Biological Sex Mismatch: Individuals whose self-identified gender does not align with their biological sex are excluded, to maintain consistency in data affected by sexual dimorphism.

Training Level: Recreational athletes, individuals with less than 3 years of high-level training, or those lacking competitive experience are excluded.

Health Conditions: Individuals with any medical conditions, chronic illnesses, acute injuries, or undergoing treatments that may interfere with athletic performance or study variables are excluded.

Medication: Use of medications or supplements that could influence metabolism, muscle composition, or overall physical performance results in exclusion.

Other Factors: Any other factors, such as lifestyle habits (e.g., smoking, excessive alcohol use), that could affect physiological responses to training and testing, are grounds for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility to participate in the study is restricted to individuals whose self-identified gender aligns with their biological sex due to the influence of sexual dimorphism on study outcomes. This alignment ensures that the physiological differences inherent between male and female bodies-such as muscle composition, metabolic rates, and hormonal profiles-are appropriately accounted for, especially in a high-performance athletic context where these factors significantly impact performance and recovery.
Study Population: The study will be conducted at the Olympic Preparation Center COS OPO in Wałcz. Testing will begin in the morning with fasting body composition measurements and blood sampling to determine baseline values of measured parameters. Psychological assessments, including questionnaires tailored for the study, will also be administered. Following this, participants will undergo an exercise test in a specialized training room equipped with modern rowing ergometers, during which each athlete will row a distance of 6,000 meters as quickly as possible. Athletes will be encouraged to maximize their effort throughout the test. Additional blood samples will be collected according to the testing schedule. The blood samples will then be transported to the ZWKF AWF laboratory in Poznań for parameter analysis.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in cortisol level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery.
  Marker of stress level.
Changes from baseline in testosterone level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery.
  Marker of anabolic activity.
Changes from baseline in serotonin level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery.
  Marker of mood regulation and emotional well-being
Changes from in serotonin level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery.
  Marker of mood regulation and emotional well-being.
Changes from baseline in gamma-aminobutyric acid (GABA) level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery.
  Marker of neuroinhibition.
Changes from baseline in dopamine level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery.
  Marker of stress and adrenal function.
Changes from baseline in tryptophan level. | At rest (before the exercise test), 1 minute after the end of the test, after 1 hour of recovery.
  Marker of mood regulation, serotonin synthesis.
Baseline Mood Profile of Athletes Before Exercise Test Using POMS Questionnaire. | At rest (before the exercise test).
  The Profile of Mood States (POMS) questionnaire measures mood states and emotional well-being.
Baseline Stress and Recovery Profile of Athletes Before Exercise Test Using RESTQ-76 Sport Questionnaire. | At rest (before the exercise test).
  The Recovery-Stress Questionnaire for Athletes (RESTQ-76 SPORT), 76-item version questionnaire measures stress and recovery balance in athletes.
Baseline Psychological Strain Assessment of Athletes Before Exercise Test Using APSQ Questionnaire. | At rest (before the exercise test).
  The Athlete Psychological Strain Questionnaire (APSQ) measures psychological strain and mental health challenges in athletes.
Baseline Eating Behavior and Attitudes of Athletes Before Exercise Test Using EDE-Q 6.0 Questionnaire. | At rest (before the exercise test).
  The Eating Disorder Examination Questionnaire (EDE-Q 6.0) measures the severity of eating disorder behaviors and attitudes.
Baseline Eating Behavior and Attitudes of Athletes Before Exercise Test Using EDE-Q 6.0 Questionnaire. | At rest (before the exercise test).
  The Eating Disorder Examination Questionnaire (EDE-Q) measures the severity of eating disorder behaviors and attitudes.
Baseline Energy Availability and Health Assessment of Female Athletes Before Exercise Test Using LEAF Questionnaire. | At rest (before the exercise test).
  The Eating Disorder Examination Questionnaire (EDE-Q) measures the severity of eating disorder behaviors and attitudes.
Baseline Energy Availability and Health Assessment of Male Athletes Before Exercise Test Using LEAM Questionnaire. | At rest (before the exercise test).
  The Eating Disorder Examination Questionnaire (EDE-Q) measures the severity of eating disorder behaviors and attitudes.

SECONDARY OUTCOMES:
Baseline Dietary Habits Assessment of Athletes Before Exercise Test Using Nutrition Questionnaire | At rest (before the exercise test).
  The nutrition questionnaire assesses dietary habits, nutrient intake, meal frequency and types, potential deficiencies or excesses, food preferences, supplement use, and overall diet quality.
Baseline Body Composition Assessment of Athletes Before Exercise Test | At rest (before the exercise test).
  Baseline body composition measurements will be conducted using the bioimpedance method to assess athletes' body fat, muscle mass, and overall composition prior to the exercise test.

CONTACTS AND LOCATIONS:
Locations (1):
- Poznań University of Physical Education, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available because protecting participant confidentiality is a priority, especially given the sensitive nature of personal health and performance data collected in this study. Additionally, there may be limitations in data-sharing infrastructure and resources needed to anonymize and securely manage IPD for external access. Ensuring compliance with privacy regulations and ethical standards also restricts the feasibility of making IPD broadly available to other researchers.